CLINICAL TRIAL: NCT05722132
Title: Latinos Kick Buts: Mobile Engagement and Cessation Support for Latinos Who Smoke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Paula Cupertino, Professor, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007635; R42MD010318 (NIH)
Record Dates: First submitted 2022-12-16; First posted 2023-02-10 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- One cycle-no monetary incentive (Active Comparator)
  Interventions: Behavioral: One cycle
- One cycle-fixed amount of incentive (Active Comparator)
  Interventions: Behavioral: One cycle; Behavioral: 5 Dollar Incentive
- One cycle-raffle as incentive (Active Comparator)
  Interventions: Behavioral: One cycle; Behavioral: Raffle Incentive
- 4 cycles- no monetary incentive (Active Comparator)
  Interventions: Behavioral: 4 cycles
- 4 cycles- fixed amount of incentive (Active Comparator)
  Interventions: Behavioral: 4 cycles; Behavioral: 5 Dollar Incentive
- 4 cycles- raffle as incentive (Active Comparator)
  Interventions: Behavioral: 4 cycles; Behavioral: Raffle Incentive

INTERVENTIONS:
Behavioral: One cycle — Message Design Participants will receive 3 messages per cycle that contain information on how to enroll in a cessation program.
  Arms: One cycle-fixed amount of incentive; One cycle-no monetary incentive; One cycle-raffle as incentive
Behavioral: 4 cycles — Participants will receive 3 messages per cycle that contain information on how to enroll in a cessation program.
  Arms: 4 cycles- fixed amount of incentive; 4 cycles- no monetary incentive; 4 cycles- raffle as incentive
Behavioral: 5 Dollar Incentive — Participants will receive 3 messages per cycle that contain information on how to enroll in a cessation program. The introductory message will mention that participants will receive $5 if they enroll in the program or that they should look out for messages with a "$" sign at the beginning that will provide an incentive if they respond.
  Arms: 4 cycles- fixed amount of incentive; One cycle-fixed amount of incentive
Behavioral: Raffle Incentive — The incentive message (indicated with a leading "$" sign) will invite participants to respond, and participants that do so will be included in a random drawing depending on the condition. The incentive message for the opportunity to win will contain a link to a website that provides full details of the timing of the drawing, the chances of winning, and when notification of winners will be made.
  Arms: 4 cycles- raffle as incentive; One cycle-raffle as incentive

SUMMARY:
Latino Kick Buts (LKB) is a smoking cessation treatment program available to Strong Memorial Hospital patients who smoke. LKB encompasses two integrated components: (1) a 12-week text messaging counseling program with interactive capabilities and (2) pharmacotherapy support (provision of nicotine replacement therapy at no cost). LKB utilization among Latinos who smoke remains minimal. This study aims to identify the types of text messages more effective in enrolling Latinos who smoke, identified in the electronic medical record, into LKB.

ELIGIBILITY:
Inclusion Criteria:

* Adult Latinos who smoke and have received medical care at Strong Memorial Hospital/SHARP healthcare within the last year.
* having smoking status recorded in the EMR

Exclusion Criteria:

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2826 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participant who enroll in cessation program | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cartujano-Barrera F, Catley D, Chavez-Iniguez A, Fox AT, Yang H, Rieth KK, Holland A, Richter K, Sherman SE, Slagle G, Werntz S, Cupertino AP. Evaluating text messaging approaches to promote enrollment in smoking cessation treatment among Latino adults: A pragmatic randomized clinical trial. Chest. 2026 Jan 10:S0012-3692(26)00009-7. doi: 10.1016/j.chest.2025.11.054. Online ahead of print. PMID 41525889